CLINICAL TRIAL: NCT03316703
Title: Surgical Treatment of the Thoracolumbar Spine Fractures - Conventional Open Surgery Versus Minimally Invasive Percutaneous Surgery: A Randomized Trial.
Brief Title: Surgical Treatment of the Thoracolumbar Spine Fractures.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Helton Defino, PhD in Orthopedics and Traumatology, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Thoracolumbar Spine Surgery
Record Dates: First submitted 2017-05-19; First posted 2017-10-20 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Spinal Fracture; Traumatic Fracture
Keywords: Spine, Spinal injuries, Fractures, Bone
MeSH Terms: conditions — Spinal Fractures; Spinal Injuries; Fractures, Bone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional open surgery (Active Comparator): Fixation of a proximal vertebra, a vertebra distal to the fractured vertebra, and also of the fractured vertebra with a pedicle fixation system using the conventional open to implant placement without subsequent arthrodesis.
  Interventions: Procedure: Conventional open surgery
- Minimally invasive percutaneous surgery (Experimental): Fixation of a proximal vertebra, a vertebra distal to the fractured vertebra, and also of the fractured vertebra with a pedicle fixation system using the percutaneous minimally invasive approach to implant placement without subsequent arthrodesis.
  Interventions: Procedure: Minimally invasive percutaneous surgery

INTERVENTIONS:
Procedure: Conventional open surgery — Surgical treatment will be performed by stabilizing the fractured vertebral segment (proximal vertebra and vertebra distal to fractured vertebra and fractured vertebra) by means of a 6.5 mm or 6.5 mm diameter polyaxial pedicle screw system. In the fractured proximal and distal vertebrae to the vertebrae, screws will be used up to the vertebral body and fractured vertebra will use shorter screws that do not penetrate the vertebral body. In the fractured vertebra, single or bilateral pedicle screw will be used according to the degree of involvement of the pedicle of the fractured vertebra.
  The vertebral fixation system will be applied through the conventional open approach (group A).
  Arms: Conventional open surgery
Procedure: Minimally invasive percutaneous surgery — Surgical treatment will be performed by stabilizing the fractured vertebral segment (proximal vertebra and vertebra distal to fractured vertebra and fractured vertebra) by means of a 6.5 mm or 6.5 mm diameter polyaxial pedicle screw system. In the fractured proximal and distal vertebrae to the vertebrae, screws will be used up to the vertebral body and fractured vertebra will use shorter screws that do not penetrate the vertebral body. In the fractured vertebra, single or bilateral pedicle screw will be used according to the degree of involvement of the pedicle of the fractured vertebra.
  The vertebral fixation system will be applied through the minimally invasive percutaneous approach (group B) according to allocation after randomization.
  Arms: Minimally invasive percutaneous surgery

SUMMARY:
The thoracolumbar segment fractures are the most frequent along the spine, and surgical treatment is indicated in unstable fractures. Surgical treatment has been performed through the posterior fixation pedicle fixation systems, and where necessary complemented by decompression of the spinal arthrodesis and previous channel. Surgical treatment has been performed by conventional open approach through the posterior incision on the midline, and detachment and removal of paraspinal muscles to access the posterior vertebral elements. The percutaneous minimally invasive surgery was introduced in the context of spinal surgery to reduce the morbidity associated with conventional open approach. It has been reported the lowest bleeding intra- and postoperative period, less pain, shorter hospital stay, rehabilitation and return to work faster with less use of minimally invasive percutaneous approach of the spine. However, predominates in the literature of clinical case reports and few prospective and randomized clinical trials. The performance of prospective randomized clinical trials have been required for the evaluation of the benefits of minimally invasive surgery in the treatment of the thoracolumbar spine fractures. The objective of the study is to compare the surgical treatment of fractures of the thoracolumbar spine using the conventional open approach or minimally invasive percutaneous approach to the stabilization of the vertebral segment affected, and using similar type of pedicle spinal fixation system. Patients will be evaluated in the preoperative, postoperative, 1,2,3,6,12 and 24 months by parameters related to the perioperative (intraoperative bleeding, surgery time), clinical (VAS, SF-36, HADS, EQ-5D-5L), images (radiographs and computed tomography). The study results will impact the guidelines of the surgical treatment of thoracolumbar spine fractures and may indicate the advantages or disadvantages of using surgery through conventional open approach to minimally invasive percutaneous surgery.

DETAILED DESCRIPTION:
Introduction: Fractures of the thoracic and lumbar spine are the most frequent fractures of the axial skeleton, and correspond to about 89% of vertebral fractures. Two-thirds of these fractures occur in the thoracolumbar transition between T11 and L2 (50% of thoracic spine fractures at T12 level and 60% of lumbar spine fractures at L1 level). Surgical treatment of thoracolumbar spine fractures has been indicated in unstable fractures with the aim of stabilizing the fractured vertebral segment and allowing early rehabilitation without the use of external immobilization and rest in the bed. Conventional surgical treatment has been performed by means of fixation and posterior arthrodesis of the vertebral segment using pedicle fixation systems with or without arthrodesis The scientific challenge of the project is to carry out this method of pioneering study in our country, as no prospective randomized clinical trial has been performed in our country to compare the outcome of surgical treatment of thoracolumbar spine fractures through conventional open surgery or surgery Minimally invasive percutaneous. There are few reports of prospective and randomized trials on this subject and its implementation has been stimulated to increase the level of evidence related to the surgical treatment of thoracolumbar spine fractures.

The objective of the study will be to compare the results of treatment of thoracolumbar spine fractures through the open approach (conventional surgery) or percutaneous (minimally invasive) approach with a pedicle fixation system without vertebral arthrodesis.

The hypothesis of the study is that minimally invasive percutaneous surgery has the advantage of producing less surgical trauma with less intra- and postoperative bleeding, lower pain intensity, shorter hospitalization time and lower rate of complications, and postero-lateral arthrodesis Is not required in the treatment of thoracolumbar spine fractures.

Material and methods

After the clinical and radiographic evaluation (simple radiographs, CT and MRI if necessary) of the patients the fracture will be classified according to the classification Magerl et al., and the therapeutic planning defined. Fractures with surgical indication by means of the posterior approach will be selected for the study and the randomization process performed individually for each type of fracture (A, B and C) according to the Magerl classification. Patients will be randomized and assigned to two groups: A - conventional open surgery and B - minimally invasive percutaneous surgery.

Surgical treatment will be performed by stabilizing the fractured vertebral segment (proximal vertebra and vertebra distal to fractured vertebra and fractured vertebra) by means of a 6.5 mm or 6.5 mm diameter polyaxial pedicle screw system. In the fractured proximal and distal vertebrae, screws will be used up to the vertebral body and in fractured vertebra shorter screws that do not penetrate the vertebral body will be used. In the fractured vertebra, single or bilateral pedicle screw will be used according to the degree of involvement of the pedicle of the fractured vertebra.

The vertebral fixation system will be applied through the conventional open approach (group A) or minimally invasive percutaneous approach (group B) according to allocation after randomization.

Patients will be evaluated through perioperative, clinical, and radiographic parameters.

Perioperative parameters:

Time of surgery - time elapsed between incision and closure of the skin. Intraoperative bleeding - a measure of the amount of blood evaluated by the amount of blood drawn and blood from the compresses and gauzes used.

Postoperative bleeding - a measure of the amount of blood aspirated through the drain and measured in the postoperative gauze pads and dressings.

Time of use of fluoroscopy. Postoperative walking time Length of hospital stay Drugs used in the postoperative period

Clinical parameters:

Visual pain scale (VAS) - evaluated in the preoperative period, 1,2,3,4,5,6,7 postoperative days, 1,2,3,6,12 and 24 months.

Medical Outcomes Study 36 - Item Short - Form Health Survey (SF-36) HADS - Hospital Anxiety Depression Scale EQ-5D-5L Dennis Pain and Work Scale Pain Assessment Scale (Dennis) P1: absence of pain P2: minimal occasional pain; No need for medication. P3: Moderate pain, occasional medication and no interruption of professional or daily activities.

P4: moderate or severe pain, occasional absence of work, significant change in daily activities.

P5: constant, severe pain, use of chronic analgesic medication

Work ability assessment scale (Dennis) W1: return to previous work (heavy arm activity) or heavy physical activities W2: return to previous work (sedentary) or heavy physical labor with restrictions W3: unable to return previous plus works full time in another activity W4: unable to return full time to work W5: does not work, totally disabled They were evaluated in the immediate postoperative period, 1,2,3,6,12 and 24 months.

Radiographic Parameters Simple radiographs in AP and profile - location, fracture classification, assessment of vertebral body height, evaluation of Farcy's sagittal index, fractured kyphosis, fractured vertebral kyphosis, intervertebral disc height above and below fractured vertebra, alignment in AP, (preoperative, immediate postoperative, 1,2,3,6,12 and 24 months).

Alignment in the coronal plane will be performed by measuring the angle of Cobb between the line parallel to the proximal vertebral plaque of the vertebra above the fractured vertebra and distal vertebral plate below the fractured vertebra.

The height of the vertebral body will be evaluated by means of the percentage of compression of the vertebral body in relation to the adjacent segments. The height of the vertebral body above (V1) and below (V2) of the fractured vertebra (V3) is considered using the following formula:% compression = [(A1 + A3) / 2-A2] / (A1 + A3) / 2

The kyphosis of the fractured segment will be assessed by the angle formed by the line parallel to the superior vertebral plate of the vertebra proximal to the fractured vertebra and by the line of the inferior vertebral plate of the vertebra distal to the fractured vertebra The sagittal index of the fractured segment (Farcy Index) will be calculated using the height of the proximal vertebra (A1), height of the fractured vertebra (A2) and height of the distal vertebra. Sagittal index of the fractured segment = (A3): 100- (2xA2 / A1 + A3) x100.

Computed tomography - morphology and type of fracture, percentage of compression of the vertebral canal, positioning of the screws (preoperative and immediate postoperative).

Compression of the vertebral canal will be evaluated by measuring the sagittal diameter of the vertebral canal (Fig. 8) and the direct measurement of the cross-sectional area of the vertebral canal using scanning to delimit its perimeter.

The positioning of the screws inside the pedicles will be evaluated by means of tomographic cuts of 2mm. Correct positioning will be considered when the pedicle screw is fully encircled by the vertebral pedicle and the cortical vertebra is not perforated. The perforation will be classified as small (≤2mm), medium (2.1-4mm) and severe (> 4mm), and the perforation site: medial, lateral, superior, posterior will also be evaluated.

Evaluation of implant release, implant breakage and fracture consolidation, loss of reduction.

Computed tomography - evaluation of the paravertebral musculature - Evaluation of the transverse sectional area and fat infiltration in the paravertebral musculature by computed tomography (CT).

The CT examinations performed to evaluate the position of the metallic implants, fracture type and the evolution of the morphology of the vertebral body will also be used to evaluate the paravertebral musculature. In this way it will be possible to compare the effect of each of the fixation techniques on the musculature trophism.

The evaluation will be performed by a senior radiologist with more than fifteen years of experience in musculoskeletal radiology and with experience in evaluation using quantitative techniques.

Patient images will be anonymized and presented to the radiologist through the Osirix imaging software at random. The observer will not be aware of the clinical and surgical information at the time of the measurements to be performed.

Two other researchers, a radiologist and a spine surgeon will perform this classification independently, so as to enable the analysis of Interobserver reproducibility of the classification.

General risks, local and adverse effects - risks will be defined as any incident, change in treatment or normal progress regardless of whether or not it is associated with the treatment being evaluated. The predicted risks related to thoracolumbar spine fractures and their surgical treatment are superficial infection, deep infection, epidural hematoma, duramater injury, inadequate position of pedicle screws, radiculopathy, fractured vertebral segment kyphosis, instability, pain uncontrollable to treatment , Failure of implants, degeneration of adjacent segments, pressure ulcers and reoperation.

The adverse effects will be considered as any undesirable medical event that the study participant presents (death, deep venous thrombosis, septicemia, pulmonary embolism, pneumonia, urinary tract infection, acute respiratory failure, multiple organ failures, hospitalization, prolonged failure of the implants Or intraoperative adverse effects).

ELIGIBILITY:
Inclusion Criteria:

* Single level fracture
* Fracture T11-L5
* Posterior Stabilization Indication

Exclusion Criteria:

* Fracture in more than 1 level
* Osteoporotic fracture
* Pathological fracture
* Previous history of surgery
* Deformity
* Mental disease
* TCE
* Posterior vertebral canal open decompression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-12-10 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | up to 24 months
  The intensity of pain will be measured by Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
Postoperative complications | immediate postoperative, and 1,2,3,6,12 and 24 months of followup
  To evaluate the rate of postoperative complications such as superficial infection, deep infection, nerve injury, vascular injury, hematoma
Postoperative adverse events | immediate postoperative, and 1,2,3,6,12 and 24 months of followup
  The adverse effects will be considered as any undesirable medical event that the study participant presents (death, deep venous thrombosis, septicemia, pulmonary embolism, pneumonia, urinary tract infection, acute respiratory failure, multiple organ failure, hospitalization, prolonged failure of the implants or intraoperative adverse effects).
Breakage or release of implants through radiographs | immediate postoperative, and 1,2,3,6,12 and 24 months of followup
  Evaluation of implant release
Breakage or release of implants through CT scan | immediate postoperative, and 1,2,3,6,12 and 24 months of followup
  Evaluation of implant release
Total costs | 24 months
  The incremental budgetary impact (IO inc) [(NiND x CtND) - (NiDA x CtDA), where NIND = number of patients under percutaneous approach; CtND = total cost of percutaneous approach; NiDA = number of patients in conventional surgery; CtDA =. Total cost of conventional approach.
Intraoperative bleeding (ml) | 48 hours postoperative
  Intraoperative bleeding - a measure of the amount of blood evaluated by the amount of blood drawn and blood from the compresses and gauzes used.
Postoperative bleeding (ml) | 48 hours postoperative
  Postoperative bleeding - a measure of the amount of blood aspirated through the drain and measured in the postoperative gauze pads and dressings.
Surgery time (in minutes) | Intraoperative
  Time of surgery - time elapsed between incision and closure of the skin.
Length of hospital stay (in days) | At discharge (up to two week post-surgery)
  Number of days stayed in hospital
Short Form Health Survey (SF-36) | 1,2,3,6,12 and 24 months.
  Patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Scores range from 0 - 100. The lower the score the more disability, while the higher the score the less disability.
Hospital Anxiety Depression Scale (HADS) | 1,2,3,6,12 and 24 months.
  Self-rating scale that measures anxiety and depression. The HADS aims to measure symptoms of anxiety and depression and consists of 14 items, seven items for the anxiety subscale (HADS Anxiety) and seven for the depression subscale (HADS Depression). Each item is scored on a response-scale with four alternatives ranging between 0 and 3. All answered are summed to obtain the two subscales. Cut-off scores are 8-10 for doubtful cases and ≥11 for definite cases.
EuroQol five-dimensional questionnaire (EQ-5D-5L) | 1,2,3,6,12 and 24 months.
  Quality of life measure. The EQ-5D-5L has five domain scales (mobility, self-care, usual activities, pain and discomfort, and anxiety and depression) and five levels for each domain. Level 1 response represents "no problems," level 2 "slight problems," level 3 "moderate problems," level 4 "severe problems," and level 5 "extreme problems" or "unable to perform," which is the worst response in the dimension. Also, respondents rate their health on a visual analogue scale ranging from 0 (the worst health imaginable) to 100 (the best health imaginable).
Vertebral segment kyphosis | preoperative, immediate postoperative, and 1,2,3,6,12 and 24 months of followup
  The kyphosis of the fractured segment will be assessed by the angle formed by the line parallel to the superior vertebral plate of the vertebra proximal to the fractured vertebra and by the line of the inferior vertebral plate of the vertebra distal to the fractured vertebra. The kyphosis of the fractured vertebra will be assessed by the angle formed by the line parallel to the upper and lower vertebral plate of the fractured vertebra using radiographs and computed tomography.
Fractured vertebral body height | preoperative, immediate postoperative, and 1,2,3,6,12 and 24 months of followup
  The height of the vertebral body will be evaluated by means of the percentage of compression of the vertebral body in relation to the adjacent segments using radiographs and computed tomography. The height of the vertebral body above (V1) and below (V2) of the fractured vertebra (V3) is considered using the following formula:% compression = [(A1 + A3) / 2-A2] / (A1 + A3) / 2
Compression of the vertebral canal | preoperative, immediate postoperative, and 1,2,3,6,12 and 24 months of followup
  Compression of the vertebral canal will be evaluated by measuring the sagittal diameter of the vertebral canal and the direct measurement of the cross-sectional area of the vertebral canal using scanning to delimit its perimeter. The sagittal diameter of the vertebral canal was defined as the distance between the posterior and anterior border of the vertebral canal.
Accuracy of the pedicle screws | preoperative, immediate postoperative, and 1,2,3,6,12 and 24 months of followup
  The positioning of the screws inside the pedicles will be evaluated by means of tomographic cuts of 2mm. Correct positioning will be considered when the pedicle screw is fully encircled by the vertebral pedicle and the cortical vertebra is not perforated.
Intraoperative fluoroscopy time (in minutes) | Intraoperative
  Time of use of fluoroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Helton LA Defino, MD, PhD., Principal Investigator — Department of Orthopedics and Traumatology.University of Sao Paulo
Locations (1):
- Hospital das Clinicas.University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Defino HLA, Costa HRT, Nunes AA, Nogueira Barbosa M, Romero V. Open versus minimally invasive percutaneous surgery for surgical treatment of thoracolumbar spine fractures- a multicenter randomized controlled trial: study protocol. BMC Musculoskelet Disord. 2019 Aug 31;20(1):397. doi: 10.1186/s12891-019-2763-1. PMID 31472691
- See also: Open versus minimally invasive percutaneous surgery for surgical treatment of thoracolumbar spine fractures- a multicenter randomized controlled trial: study protocol — http://doi.org/10.1186/s12891-019-2763-1